CLINICAL TRIAL: NCT00773292
Title: The HAM Ciclosporin Study : an Observational Trial of Therapy in Early or Progressing HAM/TSP
Brief Title: Ciclosporin in HTLV-1 Associated Myelopathy/ Tropical Spastic Paraparesis (HAM/TSP)
Acronym: HAM05
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government); University Hospital Birmingham (Other); Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cro423
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Results first posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: HTLV I Associated Myelopathy
Keywords: HAM/TSP
MeSH Terms: conditions — Paraparesis, Tropical Spastic | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ciclosporin (Experimental): 48 weeks treatment with ciclosporin
  Interventions: Drug: ciclosporin

INTERVENTIONS:
Drug: ciclosporin — Ciclosporin 2.5 - 5mg/kg/day in two equally divided doses. dose adjusted according to trough ciclosporin concentration

SUMMARY:
HAM/TSP is a chronic disease of the spinal cord, caused by a virus called HTLV-I. Worldwide approximately 20 million persons are infected.Infection with HTLV-I is lifelong, and about 3% of infected persons will develop this chronic debilitating disease, of which half will become wheelchair dependent. We, and others, have shown a strong and persistent immune response to HTLV-I in carriers and patients with HAM/TSP, but this fails to clear the virus. However, carriers with a low burden of virus in the blood have a low risk of developing disease. The immune response in these carriers seems better able to kill infected cells. A less efficient response is associated with a higher viral burden that drives the immune response with a resultant release of chemicals by the immune cells that inadvertently cause harm, most especially to cells in the spinal cord. Our understanding of HAM/TSP suggests that targeting the immune response should improve the health of our patients especially if the disease is diagnosed early. To identify the best type of treatment we are planning a series of studies of drugs that target the immune response in different ways. Each has been used in other inflammatory conditions but never before studied in HAM/TSP. We aim to study the extent and duration of the clinical response and to associate this with the different effects that the therapies have on the immune response and on the number of HTLV-I infected cells in the blood. This in turn will improve our knowledge and understanding of the disease and should lead to better therapy. This application is in relation to the first study - to explore that therapeutic benefit of ciclosporin in patients with HAM/TSP.

DETAILED DESCRIPTION:
This is a proof of concept, open, observational study of Ciclosporin for the treatment of HTLV-I-associated myelopathy in patients with less than 2 years disease or new evidence of progression. After two baseline assessments patients will be commenced on ciclosporin in a weight dependent dose (2.5 - 5mg/kg/day) and the dose adjusted according to plasma drug concentrations. Participants will be monitored on a further 11 occasion as per the schedule every 2 - 8 weeks (less frequent with time) by self-administered questionnaires relating to quality of life and spasticity, by regular assessment of pain, timed walk, spasticity, bladder and bowel function and by blood tests to ensure the safety of the therapy. Blood samples will also be collected, at the same time points, for investigation of the immune response to HTLV-I and the quantity and activity of the virus. At 5 key time points the participants will undergo a more detailed neurological examination, the spinal cord will be imaged by MRI before, once during (12 weeks) and at the completion of the study and the fluid that bathes the brain (CSF) will be examined before and after 12 weeks of therapy. Therapy is planned for 12 months with 6 months further follow-up but therapy will be continued or discontinued according to clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Early (less than 2 years) HAM
* Progressing (within past 3 months) HAM
* Important to study the effect of therapy on disease that is most active as most likely to detect and measure improvement

Exclusion Criteria:

* HIV infection
* Tuberculosis, strongyloidiasis or other infection related to immune compromise
* Hepatitis B & C viral infections
* Malignancy

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graham P Taylor, Principal Investigator — Imperial College London
Locations (1):
- National Centre for Human Retrovirology, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Martin F, Castro H, Gabriel C, Adonis A, Fedina A, Harrison L, Brodnicki L, Demontis MA, Babiker AG, Weber JN, Bangham CR, Taylor GP. Ciclosporin A proof of concept study in patients with active, progressive HTLV-1 associated myelopathy/tropical spastic paraparesis. PLoS Negl Trop Dis. 2012;6(6):e1675. doi: 10.1371/journal.pntd.0001675. Epub 2012 Jun 12. PMID 22720101

RESULTS

PARTICIPANT FLOW:
Period: Pre-treatment 4 Weeks
Arm/Group | Ciclosporin
Started | 7
Completed | 7
Not Completed | 0
Period: Treatment 48 Weeks
Arm/Group | Ciclosporin
Started | 7
Completed | 5 (Two patients discontinued the treatment but remained on the study)
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1
Period: Post Treatment 24 Weeks
Arm/Group | Ciclosporin
Started (Two patients discontinued the intervention but remained under follow up within the study) | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ciclosporin
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 50 [40 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Patient With Lack of Objective Clinical Improvement
Description: Lack of objective clinical improvement after three months of therapy. Objective improvement was defined as any of the following comparing baseline measurements to 12, 24 and 48 weeks: i) one point decrease in the IPEC 1 scale (Instituto de Pesquisa Clínica Evandro Chagas), ii) >30% improvement in 10 m timed walk, iii) visual analogue pain score reduced by >2 points, iv) reduction of frequency or nocturia by greater than one or reduction of residual volume by more than 10% at two consecutive visits.
  Proof of concept study and therefore outcomes report is descriptive only. No statistical test appropriate.
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ciclosporin
Number analyzed (Participants) | 7
Participants | 0

2. Secondary Outcome: Change in Timed Walk Rank Between Baseline and 12 Weeks
Description: Change in the time taken to walk 10 meters 0 - 12 weeks compared with baseline. A timed walk rank was created to take into account the use of walking aids.
  Timed walk rank was calculated by ranking the time to walk 10 meters over all patients and visits, in the following order (highest/worst score to lowest/best score): unable to walk; able to walk, but not able to complete 10 meters (ranked on distance walked and time taken); able to walk 10 meters with a bilateral aid; able to walk 10 meters with a unilateral aid; able to walk 10 meters unaided (all ranked on time taken).
  Decrease in score means improvement. All evaluable patients were ranked on the time taken. There is no specific range for the rank scores. Upper and lower limits vary with the number of participants evaluated
Time Frame: 0, 12 weeks
Measure: Mean (Standard Deviation); unit: rank
Arm/Group | Ciclosporin
Number analyzed (Participants) | 7
rank | -7 (5)
Statistical Analysis 1: Comparison: Ciclosporin; Test type: Other — change from baseline; p = 0.24, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 72 weeks
Arm/Group | Ciclosporin
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 1/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciclosporin (N=7)
tremor (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes